CLINICAL TRIAL: NCT01855607
Title: Topical Menthol for Chemotherapy Induced Peripheral Neuropathy (CIPN): A Randomized, Placebo Controlled Phase II Trial
Brief Title: Topical Menthol for the Treatment of Chemotherapy Induced Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Dawn L. Hershman, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AAAL2664
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Colon Cancer; Neuropathy
Keywords: chemotherapy induced neuropathy
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms | interventions — Menthol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- topical menthol (Experimental): Patients with neuropathic pain will receive topical menthol following or during chemotherapy for the treatment of either breast, gastrointestinal, or gynecologic cancer.
  Interventions: Drug: topical menthol
- placebo lotion (Active Comparator): Patients with neuropathic pain will receive placebo lotion following or during chemotherapy for the treatment of either breast, gastrointestinal, or gynecologic cancer.
  Interventions: Drug: placebo lotion

INTERVENTIONS:
Drug: topical menthol — 7.5% Methylsalicylate / 2% Menthol Lotion
  Other Names: RX-116
  Arms: topical menthol
Drug: placebo lotion — The control (placebo) product has same amount of Methylsalicylate (7.5%) and no menthol.
  Other Names: RX-115
  Arms: placebo lotion

SUMMARY:
Primary Objective: To assess whether six-week treatment with twice daily topical Menthol application will decrease neuropathic pain as measured by the change in Brief Pain Inventory-Short Form (BPI-SF worst pain score), following or during neoadjuvant/adjuvant chemotherapy with taxane or platinum-based regimens among breast, gastrointestinal or gynecologic cancer patients.

Secondary objectives:

* To compare change in patient-reported outcomes: overall BPI-SF scales, EORTC-CIPN20, European Organization for Research and Treatment of Cancer Chemotherapy Quality of Life Questionnaire (EORTC QLQ-C30), Patient-Reported Outcomes Measurement Information System (PROMIS-29) scores between study groups.
* To compare changes in dose delivery and early treatment discontinuation rates between study groups.
* To compare objective sensory and motor functional change from baseline with the use of quantitative neurosensory testing.
* To perform an exploratory analysis evaluating the interaction between treatment and chemotherapy type.

DETAILED DESCRIPTION:
Chemotherapy induced peripheral neuropathy (CIPN): CIPN is a debilitating and often irreversible toxicity associated with various chemotherapy agents widely used in the treatment of both solid tumors and hematologic malignancies. Clinical trials with Taxane-based forms of chemotherapy, commonly used in the adjuvant treatment of breast cancer, have reported up to 33% grades 2-3 sensory neuropathy and up to 14% of motor neuropathy. Severity is closely related to chemotherapy dose and schedule. CIPN may also develop in up to 64% of patients treated with 12 cycles of Oxaliplatin based adjuvant chemotherapy, when assessed clinically and electro physiologically. Patients develop an axonal, predominately sensory peripheral neuropathy, of mild to moderate severity. Thermal hyperalgesia with cold allodynia was found to be a clinical marker of early oxaliplatin neurotoxicity and may predict severe neuropathy

ELIGIBILITY:
Inclusion Criteria:

1. Age≥21 years
2. History of stage I-III breast, gastrointestinal or gynecologic cancer
3. Must have received at least one taxane or platinum based chemotherapy drug within two years prior to enrollment.
4. Must exhibit a typical symptom of CIPN that was not present prior to chemotherapy. Symptoms include numbness, tingling, thermal hyperalgesia, cold allodynia in the hands and/or feet, muscle weakness or unsteady gait in at least two of the last seven days prior to registration.
5. Signed informed consent
6. Concomitant biologic, hormonal, or radiation therapy are acceptable
7. Narcotics, antidepressants or other medications for the treatment of CIPN are permitted, if patient on a stable dose for at least one month prior to enrollment

Exclusion Criteria:

1. Previous treatment with topical menthol (menthol/methylsalicylate products like BenGay, Aspercreme, or Icy Hot) of any concentration within the previous 3 months
2. Known diabetic neuropathy
3. Severe concomitant illnesses
4. Known allergy or preexisting skin disease which prohibits use of menthol
5. Any topical treatment for neuropathy or other serious skin condition on the hands or feet.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated before randomization could be assigned, therefore all participant data is presented as a combined total and cannot be presented per Arm.
Groups:
- All Participants: Patients with neuropathic pain will receive topical menthol or placebo lotion following or during chemotherapy for the treatment of either breast, gastrointestinal, or gynecologic cancer.
  Topical menthol: 7.5% Methylsalicylate and 2% Menthol Lotion
  Placebo lotion: 7.5% Methylsalicylate and no menthol.
Period: Overall Study
Arm/Group | All Participants
Started | 12
Completed | 0
Not Completed | 12
Not completed — Withdrawal by Subject | 1
Not completed — Study was terminated | 11

BASELINE CHARACTERISTICS:
Population: The study was terminated before randomization could be assigned, therefore all participant data is presented as a combined total and cannot be presented per Arm.
  12 participants were enrolled, and 1 withdrew consent, therefore 11 participants are presented in the Baseline Analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Brief Pain Inventory-Short Form Score
Description: The Brief Pain Inventory-Short Form (BPI-SF) is a well-validated clinical tool used frequently to assess severity of pain and its effect on daily functions in patients with neuropathy. The instrument gives several ratings of the intensity and severity of pain and the degree of pain interference on activity, mood, sleep, relations with others and work. The questionnaire uses a 0-10 scale with a higher score indicating a worse outcome.
Time Frame: Baseline and 6 weeks
Population: The study was terminated due to poor enrollment; no data was collected from participants. Participants were not randomized, therefore results are reported as a combined total and cannot be presented per Arm.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in EORTC-CIPN20 Score
Description: The European Organization for Research and Treatment of Cancer Chemotherapy-induced peripheral neuropathy (EORTC-CIPN20) is a questionnaire measuring patient reported symptoms of chemotherapy induced neuropathy. Scores range from 20-80 with a higher score indicating a worse outcome.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Sensorimotor Function
Description: Sensorimotor function as measured by a Bio-Thesiometer, which measures changes in vibratory perception. The Bio-Thesiometer is an electrical tuning fork whose amplitude can be gradually increased. Vibration threshold will be assessed at the dorsum of the distal interphalangeal joint of the index finger and dorsum of the interphalangeal joint of the hallux. Subjects will be asked to indicate when the vibration stimulus is initially felt (perception threshold) and when the stimulus disappears (disappearance threshold.) The vibration perception threshold is the average of three paired measurements.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: The study was terminated before randomization could be assigned, therefore all participant data is presented as a combined total and cannot be presented per Arm.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes